CLINICAL TRIAL: NCT05439369
Title: Natriuretic Peptides as a Prognostic and Risk Stratification Tool in Assessment of Valvular Heart Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Muhammad Khidr Ezzat thabet, Resident Doctor, Assiut University
Other Study IDs: NPs in Valvular heart diseases
Record Dates: First submitted 2022-06-17; First posted 2022-06-30 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Valvular Heart Disease Stenosis and Regurgitation
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
NPs can be used To detect subset of asymptomatic with subtle LV dysfunction for further evaluation and earlier referral for intervention and its correlation with echocardiographic finding.

DETAILED DESCRIPTION:
Each patient included in the study will undergo:

1. History taking:

   Analysis of patient symptoms and signs (dyspnea , orthopnea , Paroxysmal nocturnal dyspnea, lower limb edema , tachypalpitations,…etc )
2. Clinical examination:

   * Detecion of each patient body weight , height , calculation of BMI.
   * General examination for detection of signs of Heart failure (raised JVP , lower limb edema, ..etc)
   * Examination to respiratory system
   * Auscultation of the heart for detection of valvular affection before echocardiography

Invesigations:

Laboratory investigations:

Urea and creatinine . b) ECG : for exclusion of atrial fibrillation and other arrythmias. 2D Transthorathic Echocardiography (TTE) Evaluation of valve morphology and thickness , gradients and valve area , regurgitant lesions and its severity.

Evaluation of internal cardiac dimensions and function. 5- Natriuretic peptides: as a useful screening tool to differentiate symptomatic and asymptomatic patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients echocardiographically diagnosed with significant valve lesions. Rheumatic Heart disease with significant but asymptomatic valvular Heart Disease especially (Mitral valve disease )(MS and MR) Gender: male & female

Exclusion Criteria:

* Cases with increased level of BNP as in :

Renal impairment Advanced age and obesity Atrial fibrillation and acute coronary syndromes Prior lung diseases and acute illness

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: the study will include consecutive eligible patients recruited in assiut university hospital
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
early detection of subclinical LV dysfunction. | 1 year
  early detection of subclinical LV dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Aly Abdelhafez, Lecturer, Principal Investigator — Assiut University
Locations (1):
- Assiut University ,faculty of medicine, Asyut, Egypt